CLINICAL TRIAL: NCT02371005
Title: Oral Manifestations of Systemic Sclerosis: Toward the Identification of New Prognostic Markers
Brief Title: Oral Manifestations of Systemic Sclerosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: scleroderma patients were difficult to recruit
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 6026
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Measurement of the periodontal ligament space (Other): Evaluation of the width of the ligament in patients with SSc and comparison to the width found in control.
  Interventions: Radiation: Cone Beam Computed Tomography (CBCT)
- Radiographic analysis of oro-facial manifestations (Other): Establishment of a complete clinical phenotypic description of oral manifestations associated with SSc and comparison with the control group.
  Interventions: Radiation: Cone Beam Computed Tomography (CBCT)

INTERVENTIONS:
Radiation: Cone Beam Computed Tomography (CBCT)

SUMMARY:
Systemic sclerosis (SSc) is a rare multisystem connective-tissue disorder characterized by three major pathological hallmarks: widespread fibrosis, vasculopathy and immunological abnormalities. As all connective tissues can be affected, this condition has multiple effects on the orofacial region. Indeed, the latter is involved in approximately 80% of SSc patients. Oral manifestations have a major impact on quality of life and require specific treatments that should be performed as early as possible.

Widening of the periodontal ligament space, that seems to be linked to an increased collagen synthesis, is one of the most common dental radiographic finding. However, this radiologic sign has been mostly studied on two-dimensional radiographs. The investigators have recently described in a patient suffering from SSc the existence of calcifications within the periodontal ligament space using Cone Beam Computed Tomography (CBCT) approach (Jung et al., Oral Surg Oral Med Oral Pathol Oral Radiol 2013). Such calcifications, that have never been observed before, could be part of the phenotypic spectrum of the disease, in particular when dystrophic calcinosis is associated. They could furthermore constitute a specific feature of SSc. However, this radiographic sign requires to be investigated in a largest number of patients.

Several cytokines have been implicated in SSc pathogenesis. A recent study has revealed that elevated CXCL4 serum levels correlate with disease complications, suggesting that this molecule could be used as a prognostic biomarker. Increased IL-6 serum levels also correlate with SSc severity. Gingival crevicular fluid can be easily collected from the gingival crevice surrounding the teeth and constitute an indicator of local but also systemic inflammation. Analysis of gingival crevicular fluid cytokine profile could contribute to the identification of specific SSc biomarkers and allow a better comprehension of oral manifestations pathogenesis.

The aim of this case-control study is to characterize precisely the oral manifestations associated with SSc within the National Referral Center for Rare Autoimmune Diseases (Strasbourg, France) patient cohort in order to identify specific radiological, clinical and/or biological signs. Some of them could be correlated to the severity or to the prognosis of the disease. To the investigators knowledge it is the first study using tridimensional CBCT approach.

ELIGIBILITY:
Inclusion Criteria:

* Common inclusion criteria
* Males and females ≥ 18 years (18th birthday completed)
* Affiliation to a social security scheme
* Signed informed consent form prior to inclusion in the study
* More than 12 natural teeth suitable for evaluation

Inclusion criteria for systemic sclerosis patients

* Systemic sclerosis Inclusion criteria for control
* Subjet that underwent or must undergo an upper and a lower jaw bone Cone Beam Computed Tomography examination (impacted teeth assessment, implant treatment planning)

Exclusion Criteria:

Common exclusion criteria

* Overt acute or chronic infection (HIV, viral hepatitis…) known at the time of the oral examination
* Progressive neoplasia or neoplasia diagnosed within 2 years prior to the study
* Ongoing antibiotic treatment or within 3 months before oral examination
* Individuals at risk of infective endocarditis
* Oral antiseptics within the week before oral examination (chlorhexidine mouthwashes…)
* Periodontal specialized treatments, root scaling/root planning or periodontal surgical treatment within the year before oral examination
* Ongoing medical treatment inducing a significant modification of the gingival state (anti-epileptic drugs…)
* Smoking (≥ 10 cigarettes per day)
* Pregnancy female subjects (positive urine pregnancy test)
* Lactating female subjects
* Impossibility to provide accurate informations (emergency situation, comprehension difficulties…)

Exclusion criteria for systemic sclerosis patients

* Patient currently involved in an other clinical trial (drug) or in an exclusion period following participation in another clinical trial
* Other associated systemic auto-immune disease (Sjögren syndrome with positive serum anti-SSA and/or anti-SSB auto-antibodies, systemic lupus erythematosus…)
* Progressive chronic illness other than systemic sclerosis (diabetes…)
* Immunosuppressive therapy during the last month
* Corticosteroid ≥10 mg/day during the last month
* Hematopoietic stem cell transplant recipient
* Another cause of skin sclerosis (radiotherapy on the oro-facial region…)

Exclusion criteria for control

* Systemic chronic or evolutive illness at the time of the inclusion
* Progressive pathology involving the maxilla or the mandible at the time of the inclusion (tumor…)
* Ongoing treatment with corticsteroids or non-steroidal anti-inflammatory drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Measurement of the periodontal ligament space width at mid-root level on Cone Beam Computed Tomography (CBCT) axial views | Baseline

SECONDARY OUTCOMES:
Radiographic analysis of oro-facial manifestations associated with systemic sclerosis using high-resolution volumetric Cone Beam Computed Tomography (CBCT) exploration | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sophie JUNG, Dental surgeon, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de parodontologie, Strasbourg, France

REFERENCES:
- [Derived] Jung S, Gavriiloglou M, Severac F, Haumesser L, Sayeh A, Chatelus E, Martin T, Huck O. Influence of systemic sclerosis on periodontal health: A case-control study. J Clin Periodontol. 2023 Oct;50(10):1348-1359. doi: 10.1111/jcpe.13846. Epub 2023 Jul 11. PMID 37431838